CLINICAL TRIAL: NCT01291602
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability and Pharmacokinetics of NXL104 Alone and in Combination With Ceftazidime Administered as Single and Repeated Intravenous Doses in Healthy Japanese Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of NXL104 Alone and in Combination With Ceftazidime Administered as Single and Repeated Intravenous Doses in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4280C00010
Record Dates: First submitted 2011-02-06; First posted 2011-02-08 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy Male and Female Japanese Volunteers
Keywords: NXL104; ceftazidime; CAZ104; Healthy Japanese volunteers; Phase 1; Single and Multiple Dose Study
MeSH Terms: interventions — avibactam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NXL104 (Experimental): Six Japanese subjects to receive single and repeated 500 mg IV infusions of NXL104
  Interventions: Drug: NXL104
- Placebo (Placebo Comparator): Three Japanese subjects to receive placebo IV doses
  Interventions: Drug: Placebo
- Ceftazidime NXL104 (CAZ104) (Experimental): Six Japanese subjects to receive single and repeated IV infusions of 500 mg NXL104 with 2000 mg ceftazidime
  Interventions: Drug: CAZ104

INTERVENTIONS:
Drug: NXL104 — IV Solution
  Arms: NXL104
Drug: CAZ104 — IV Solution
  Arms: Ceftazidime NXL104 (CAZ104)
Drug: Placebo — IV saline
  Arms: Placebo

SUMMARY:
This is a single and multiple dose study in healthy male and female (of non-childbearing potential) Japanese volunteers, to assess the safety, tolerability, and blood and urine drug levels of intravenous (IV) NXL104 alone and when given in combination with ceftazidime.

ELIGIBILITY:
Inclusion Criteria:

* To be considered as 'Japanese', both of the volunteer's parents, and all grandparents must be Japanese. The volunteer must have been born in Japan, have a valid Japanese passport and must not have lived outside Japan for more than 5 years
* Have a body mass index (BMI) between 17 and 27 kg/m2 inclusive and weigh at least 45 kg and no more than 100 kg.
* Females must not be lactating, and must be of non-childbearing potential (post-menopausal at least 12 months or documented irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation

Exclusion Criteria:

* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Symptoms of a clinically significant illness in the 3 months before the study
* History of hypersensitivity (eg, anaphylaxis), serious allergy, or any serious reaction to carbapenem, cephalosporins, or other β-lactam antibiotics
* Use within 14 days prior to the first study dose of any over-the-counter (including St. John's Wort or any herbal products) or prescription medication
* Smoker of more than 5 cigarettes/day or equivalent use of nicotine products during the previous 3 months

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Adverse events will be monitored as a measure of safety and tolerability | A range of 12 days
Vital signs, physical examinations, clinical laboratory tests, 12 lead electrocardiogram (ECG) and digital ECG will be assessed as a measure of safety and tolerability | A range of 12 days

SECONDARY OUTCOMES:
The pharmacokinetic parameters of plasma of NXL104 alone or in combination with ceftazidime | Range of 8 days
The pharmacokinetic parameters of urine of NXL104 alone or in combination with ceftazidime | Range of 8 days
The level of intestinal bacterial flora of NXL104 alone or in combination with ceftazidime | Range of 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MD, Study Director — AstraZeneca; Mark Yen, MD, Principal Investigator — PAREXEL Early Phase/California Clinical Trials Medical Group
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland

REFERENCES:
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- See also: Study Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1456&filename=D4280C00010_Study_Synopsis.pdf